CLINICAL TRIAL: NCT03711071
Title: ICE - Ideas, Concerns, Expectations. Implementing Patient-centered Communication to Prevent Unnecessary Medicine
Brief Title: Ideas, Concerns, Expectations. Implementing Patient-centered Communication
Acronym: ICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); University of Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 01COM180911
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Communication; Back Pain
Keywords: patient-centered-communication; Primary Care; over investigation; communication; consultation; shared-decision making; medical education; low back pain
MeSH Terms: conditions — Communication; Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Cluster randomised parallel design: Randomization to ICE communication training will take place at the practice level with units of randomizations being single handed or group practices.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participating doctors will be blinded towards the explicit purpose and design of the study. ICE communication training will be offered to all participants: to the doctors in the intervention group as a true intervention at the beginning of the trial, and to the doctors in the control group as a pretend intervention at the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Intervention Group is allocated to a Workshop of communication training before data collection covering theoretical background and clinical implementation of ICE communication in association with frequent consultation contents.
  Interventions: Other: Workshop "ICE training"
- Control Group (No Intervention): This group will not get the intervention before data collection.

INTERVENTIONS:
Other: Workshop "ICE training" — The workshop includes training in communication skills in relation to evidence based medicine.
  Arms: Intervention Group

SUMMARY:
Exploring patients' ideas, concerns and expectation (ICE) is a communication tool to promote patient centredness and shared decision making during a consultation. This study evaluates whether offering ICE training to doctors can decrease overdiagnosis in the management of acute backache.

DETAILED DESCRIPTION:
The study is a cluster randomized trial recruiting general practitioner from practices in Northern Bavaria/Germany forming a research network within the recently implemented framework of PRO PRICARE (Preventing Overdiagnosis in Primary Care).

At baseline, the intervention group (24 out of 48 doctors) will take part in a one-day training session covering theoretical background and clinical implementation of ICE communication in association with frequent consultation contents.

Primary outcome measure are referrals to physiotherapists and medical specialists such as orthopaedic surgeons, neurologists and radiologists, obtained from routinely collected practice data. Secondary outcomes are patients' and doctors' satisfaction measured via structured questionnaires and semi-structured interviews. Blinding is attempted by hiding the trial purpose and treatment allocation from the participating doctors.

ELIGIBILITY:
Inclusion Criteria:

* aged 18
* first time seeing doctor because of the defined high frequent consultation issue referring on recommendation of the National Guideline

Exclusion Criteria:

* not first time seeing the doctor during the recommended time of the National Guideline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
number of medical referrals | data collection up to 12 weeks post intervention aims to capture 40 consultations for acute backpain
  referrals of patients to physiotherapists and medical specialists such as radiologists, neurologists, orthopedic surgeons

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kühlein, Prof. Dr., Study Chair — Institute of General Practice, Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Institute of General Practice, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schedlbauer A, Burggraf L, Hueber S, Terzakis-Snyder IA, Kuhlein T, Roos M. Referrals for uncomplicated lower back pain: a cluster parallel randomised trial of patient-centred communication to improve the management of acute back pain in primary care. A study protocol. BMJ Open. 2019 Oct 28;9(10):e027718. doi: 10.1136/bmjopen-2018-027718. PMID 31662352